CLINICAL TRIAL: NCT07009457
Title: An Open Label, Multicenter Phase I Clinical Study on the Pharmacokinetics, Safety, Tolerability, and Efficacy of SHR-1316 (SC) Combined With Carboplatin and Etoposide in First-line Treatment of Extensive Stage Small Cell Lung Cancer
Brief Title: Phase I Clinical Study of SHR-1316 (SC) Combined With Carboplatin and Etoposide as First-line Treatment for Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316(sc)-101
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Widespread Small Cell Lung Cancer
MeSH Terms: interventions — Injections; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1316 (sc) Dose A Group (Experimental)
  Interventions: Drug: SHR-1316 (sc) Injection; Drug: SHR-1316 Injection; Drug: Carboplatin Injection; Drug: Etoposide Injection
- SHR-1316 (sc) Dose B Group (Experimental)
  Interventions: Drug: SHR-1316 (sc) Injection; Drug: SHR-1316 Injection; Drug: Carboplatin Injection; Drug: Etoposide Injection
- SHR-1316 (sc) Dose C Group (Experimental)
  Interventions: Drug: SHR-1316 (sc) Injection; Drug: SHR-1316 Injection; Drug: Carboplatin Injection; Drug: Etoposide Injection

INTERVENTIONS:
Drug: SHR-1316 (sc) Injection — SHR-1316 (sc) injection.
Drug: SHR-1316 Injection — SHR-1316 injection.
Drug: Carboplatin Injection — Carboplatin injection.
Drug: Etoposide Injection — Etoposide injection.

SUMMARY:
This study is a multicenter, open label phase I clinical trial aimed at evaluating the pharmacokinetics, tolerability, safety and immunogenicity of SHR-1316 (sc) subcutaneous administration combined with carboplatin and etoposide as first-line treatment for extensive stage small cell lung cancer, and to observe the initial anti-tumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with extensive stage small cell lung cancer confirmed by histology or cytology; Has not received first-line systemic therapy or immune checkpoint inhibitor treatment for ES-SCLC in the past.
2. ECOG physical fitness score 0-1 points.
3. According to RECIST v1.1, there must be at least one measurable tumor lesion.
4. Expected survival time ≥ 12 weeks.
5. Having sufficient bone marrow and organ function.
6. Participants must give informed consent to this study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria

1. Patients with central nervous system or meningeal metastases.
2. Spinal cord compression that cannot be cured by surgery and/or radiotherapy cannot be included in the study.
3. Patients diagnosed by researchers with uncontrollable tumor related pain.
4. Symptomatic third space effusion requires repeated drainage, such as pericardial effusion, pleural effusion, and abdominal effusion that cannot be controlled by pumping or other treatments.
5. Having undergone major organ surgery (excluding biopsy) or significant trauma within 4 weeks prior to the first use of the investigational drug, or requiring elective surgery during the trial period.
6. History of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, radiation pneumonitis requiring steroid treatment, or clinically significant active pneumonia at screening; Or other moderate to severe lung diseases that seriously affect lung function (patients with a history of radiation pneumonitis (fibrosis) in the radiation area may participate in this study).
7. Severe infections, including but not limited to bacteremia requiring hospitalization and severe pneumonia, were present within 4 weeks prior to the first medication; Within 2 weeks prior to the first medication, there is an active infection with CTCAE ≥ 2 that requires treatment with systemic antibiotics.
8. Individuals with active pulmonary tuberculosis infection detected through medical history or CT examination within the year prior to enrollment, or those with a history of active pulmonary tuberculosis infection more than one year ago but without formal treatment.
9. History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplant recipients.
10. Known to have alcohol or drug dependence; Individuals with mental disorders or poor compliance; Pregnant or lactating women; Or the researcher believes that there is a history of other serious systemic diseases or other reasons that make it unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
SHR-1316 serum trough concentration (Ctrough) | Day1 pre-dose to Day28.
Area under the concentration curve from time 0 to 21 days for SHR-1316 (sc) (AUC0-21d) | Day1 pre-dose to Day21.
Area under the concentration curve from time 0 to 28 days for SHR-1316 (sc) (AUC0-28d) | Day1 pre-dose to Day28.

SECONDARY OUTCOMES:
Maximum Concentration of SHR-1316 (sc) (Cmax) | Day1 pre-dose to Day28.
Time to maximum plasma concentration (Tmax) | Day1 pre-dose to Day28.
Terminal half-life (t1/2) | Day1 pre-dose to Day28.
Incidence and severity of adverse events (AEs) | About 2 years.
Objective Response Rate (ORR) | About 2 years.
Duration of Relief (DoR) | About 1.5 years.
Disease Control Rate (DCR) | About 2 years.
Progression-free Survival (PFS) | About 2 years.
Overall Survival (OS) | About 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided